CLINICAL TRIAL: NCT06036706
Title: Neurocognitive Impact of Different Irradiation Modalities for Patients With Grade I-II Skull Base Meningioma: A Prospective Multi-Arm Cohort Study
Brief Title: Neurocognitive Impact of Different Irradiation Modalities for Patients With Grade I-II Skull Base Meningioma:
Acronym: CANCER-COG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Région Normandie (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A02097-36
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Meningioma; Radiation Toxicity
MeSH Terms: conditions — Meningioma; Radiation Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort "IMRT": (Other): Patients receiving normo-fractionated intensity-modulated brain irradiation with or without stereotactic positioning (IMRT, VMAT, Tomotherapy…)
  Interventions: Radiation: Normo-fractionated intensity-modulated brain irradiation with or without stereotactic positioning
- Cohort "SRT" (Other): Patients receiving hypo-fractionated stereotactic brain irradiation
  Interventions: Radiation: Hypo-fractionated stereotactic brain irradiation
- Cohort "PRT" (Other): Patients receiving normo-fractionated proton therapy brain irradiation
  Interventions: Radiation: Normo-fractionated proton therapy brain irradiation
- Control cohort (Other): Participants without any meningioma, cancer history or neurological comorbidities
  Interventions: Other: Cognitive assessment by a trained neuropsychologis

INTERVENTIONS:
Radiation: Normo-fractionated intensity-modulated brain irradiation with or without stereotactic positioning — Patients receiving normo-fractionated intensity-modulated brain irradiation with or without stereotactic positioning (IMRT, VMAT, Tomotherapy…)
  Arms: Cohort "IMRT":
Radiation: Hypo-fractionated stereotactic brain irradiation — Patients receiving hypo-fractionated stereotactic brain irradiation
  Arms: Cohort "SRT"
Radiation: Normo-fractionated proton therapy brain irradiation — Patients receiving normo-fractionated proton therapy brain irradiation
  Arms: Cohort "PRT"
Other: Cognitive assessment by a trained neuropsychologis — Participants without any meningioma, cancer history or neurological comorbidities will undergo cognitive assessment by a trained neuropsychologist, similarly as for patients
  Arms: Control cohort

SUMMARY:
For the purpose of this research, investigator will constitute several cohorts of patients, treated either by intensity-modulated radiotherapy, stereotactic radiotherapy or proton-therapy. This will allow better understanding the cognitive and anatomical damages caused by new radiotherapy techniques and better understanding how ionising radiation (X-rays or protons) acts in the long term on brain tissue. Longitudinal follow-up will be multimodal, based on yearly multi-parametric brain MRI to assess morphological changes, in relation with dosimetric data as well as neuropsychological performances, health-related quality of life, anxiety and depression disorders, memory tasks, and socio-professional reintegration. This will notably make it possible to evaluate the relationship between dosimetric data, age at the time of treatment, region of the brain irradiated, type of radiation used, dose per fraction, neurocognitive and neuro-anatomical consequences. A Normal Tissue Control Probability (NTCP) model will be also developed. Overall, the results of this study should contribute to the improvement of treatment techniques, in particular by preserving as much as possible the significant cerebral zones (hippocampi, frontal lobe, sub-ventricular zones, etc.), and to the management of patients by proposing appropriate support measures. In the proton-therapy cohort, evaluations will make it possible to establish more precisely the place that this new irradiation strategy should occupy in the management of low grade meningioma. Importantly, investigator have planned to constitute a last cohort, with subjects free of any neurological disease, to make it easier the interpretation of cognitive performances over time among patients in the three brain radiation cohorts.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Benign meningioma (grade I), or atypical meningioma (grade II)
* Histologic proven of benign meningioma, atypical meningioma or unequivocal radiological diagnosis of skull base meningioma if biopsy is recused.
* Indication of irradiation validated by a multidisciplinary meeting
* Age >20 years and <65 years
* Expected overall survival >10 years
* Adjuvant or exclusive irradiation is allowed.
* Signed informed consent form
* WHO Performance status equal to 0 or 1
* Patient affiliated to the French social health insurance
* Patient whose neuropsychological abilities allow to follow the requirements of the protocol

Exclusion Criteria:

* Patient with mutation in a known predisposition gene (NF-2, SMARCE-1).
* Cerebrovascular pathology, presence of other tumors of the nervous system, congenital malformations of the nervous system, multiple sclerosis, Parkinson's disease, organic psychosis (other than dementia), or schizophrenia.
* Other localization than skull base meningioma
* Histology/radiological features rather different than grade I-II meningioma
* Histologic proven grade III meningioma
* Uncontrolled epilepsy
* Contraindication to MRI
* Patient with a history of brain irradiation.
* Patient with a history of cancer in the last five years (excluding skin baso-cellular carcinoma)
* Pregnant/breastfeeding woman
* Any geographical conditions, social and associated psychopathology that may compromise the patient's ability to participate in the study
* Participation in a therapeutic trial evaluating a radiotherapy schedule or a new drug or combination for less than 30 days
* Patient deprived of freedom or under guardianship
* Hypersensibility to Gadolinium

Participants free of brain disease or cancer history:

Inclusion Criteria:

* Subject without any history of neurological disease (cerebral stroke, epilepsy, Intra cranial Neurosurgery procedure, meningioma, pituitary adenoma, Parkinson disease,Dementia…) or absence of personality disorders and progressive psychiatric pathology
* Age >20 years and <65 years
* Signed informed consent form
* WHO Performance status equal to 0 or 1
* Subject affiliated to the French social health insurance
* Subject whose neuropsychological abilities allow to follow the requirements of the protocol
* No major cognitive disorder that may compromise the realization of cognitive evaluations, defined as a MoCA score in accordance with the threshold depending on age and educational level according to the GRECOGVASC normative data

Non-inclusion criteria

* Cerebrovascular pathology, presence of other tumors of the nervous system, congenital malformations of the nervous system, multiple sclerosis, Parkinson's disease, organic psychosis (other than dementia), or schizophrenia
* History of epilepsy with antiepileptic drug
* Subject with a history of brain irradiation
* Subject with a history of cancer in the last five years (Excluding skin baso-cellular carcinoma)
* Pregnant/breastfeeding woman
* Any geographical conditions, social and associated psychopathology that may compromise the subject's ability to participate in the study
* Participation in a therapeutic trial - Subject deprived of freedom or under guardianship

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2038-09 (Estimated); Study Completion 2039-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of cognitive impairment (a total of ≥ 5 impaired z-scores) | 10 years
  Occurrence of cognitive impairment in comparison with baseline evaluation (before brain irradiation), evaluated with z-scores

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - centre François Baclesse, Caen
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Henri Becquerel, Rouen

REFERENCES:
- [Derived] Lesueur P, Joly F, Clarisse B, Lequesne J, Stefan D, Balosso J, Lange M, Thureau S, Capel A, Castera M, Legrand B, Goliot N, Grellard JM, Tessonnier T, Castel H, Valable S. Neurocognitive impact of different irradiation modalities for patients with grade I-II skull base meningioma: a prospective multi-arm cohort study (CANCER COG). Radiat Oncol. 2025 Jan 29;20(1):16. doi: 10.1186/s13014-025-02591-1. PMID 39881369